CLINICAL TRIAL: NCT00203710
Title: A Single-Center Controlled Registry to Evaluate the Concentric Retriever System for the Treatment of Stroke
Brief Title: Concentric Retriever Device (CRD) in Acute Ischemic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Starkman (Other)
Responsible Party: Sponsor-Investigator, Sidney Starkman, Clinical Professor, Emergency Medicine and Neurology, University of California, Los Angeles
Organization: University of California, Los Angeles (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCLA-TR-001
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Acute Ischemic Stroke
Keywords: Concentric Retriever Device; embolectomy; acute ischemic stroke; treatment
MeSH Terms: conditions — Ischemic Stroke

INTERVENTIONS:
Device: Concentric Retriever Device

SUMMARY:
The primary purpose is to study the safety and effectiveness of the Concentric Retriever Device(CRD)in ischemic stroke patients who undergo clot retrieval with the CRD within 8 hours of stroke symptom onset. The CRD has been approved by the U.S. Food and Drug Administration to retrieve foreign bodies (such as pieces of metal) from blood vessels in the body. The CRD is a small metal wire with a loop at the end (like a corkscrew) that removes clots from arteries and thereby restores blood flow to the brain. Prior versions of the CRD may have been too soft to pull out clots, just as a corkscrew that is too soft would not pull out corks. The current version of the CRD is not as soft and may be more effective in retrieving clots. Hypothesis: By restoring blood flow to the brain, stroke symptoms may get better or the stroke may be prevented from getting worse.

DETAILED DESCRIPTION:
The primary objective is to assess the safety and efficacy of the Concentric Retriever in the treatment of thrombotic occlusions originating in the internal carotid, middle cerebral (M1 and M2 segments), basilar, posterior cerebral or vertebral arteries. A maximum of 50 patients may be enrolled at a single site, University of California, Los Angeles.

Primary endpoints: Achievement of recanalization (TIMI/TICI grade II or III flow) immediately post procedure without occurrence of major complications will be assessed. Major complications are defined as vessel perforation, intramural arterial dissection, symptomatic intra-cranial hemorrhage, and significant embolization in a previously uninvolved arterial territory.

Secondary endpoints: Assessment of patient's neurological condition and functional state using the NIHSS, Barthel Index, and Modified Rankin at 30 and 90 days post-procedure. A composite of major adverse events at 30 and 90 days post-procedure will be reported. Major adverse events are defined as death and new stroke.

ELIGIBILITY:
Inclusion Criteria:

1(a) -Patients who present within 8 hours of stroke onset and are not candidates for treatment with t-PA who have clinical signs consistent with the diagnosis of ischemic stroke such as impairment of language, motor function, sensation, cognition, and/or gaze, or vision.

1(b). Patients who have had an acute ischemic stroke treated with intravenous thrombolytic therapy where vascular imaging (TCD, CTA, MRA, angiography) shows a persistent occlusion after the end of the infusion treatment.

2. Patients > 18 years of age. 3. NIHSSS > 7 4. Angiogram shows a thrombotic occlusion originating in the internal carotid, middle cerebral (M1 or M2 segment), basilar, posterior cerebral, or vertebral arteries.

5. Patient/patient guardian is willing to comply with the protocol requirements and return to the treatment center for all required clinical evaluations.

Exclusion Criteria:

1. Patient is pregnant (if within child bearing age).
2. Patient has baseline glucose of < 50mg/dL (<50 mg/mM).
3. Patient has excessive arterial tortuosity that precludes the device from reaching the target area.
4. Patient has known hemorrhagic diathesis, coagulation factor deficiency, or oral anticoagulant therapy with INR > 2.0.
5. Patient received Heparin within 48 hours with a PTT greater than 2 times the lab normal.
6. Patient has baseline platelets < 30,000.
7. Patient has history of severe allergy to intra-arterial contrast medium.
8. Patient has severe, sustained hypertension (systolic blood pressure > 185 mm Hg or diastolic blood pressure > 110 mm Hg).

   NOTE: If the blood pressure can be successfully reduced and maintained at the acceptable level using medication (i.e. Nipride), the patient can be enrolled.
9. CT Scan or MRI reveals significant mass effect with midline shift.
10. Patient's angiogram shows an arterial stenosis (>50%) proximal to the embolus.
11. Patient's anticipated life expectancy is less than 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2003-10; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Achievement of recanalization (TIMI/TICI grade II or III flow) immediately post procedure.
In addition, major complications defined as vessel perforation, intramural arterial dissection, symptomatic intra-cranial hemorrhage, and significant embolization in a previously uninvolved arterial territory will be tabulated.

SECONDARY OUTCOMES:
Assessment of patient's neurological condition and functional state using the NIHSS, Barthel Index, and
Modified Rankin at 30 and 90 days post-procedure.
A composite of major adverse events at 30 and 90 days post-procedure. Major adverse events are defined as death and new stroke.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States